CLINICAL TRIAL: NCT04381897
Title: Use of N-Acetylcysteine (NAC) in the Treatment of Repetitive Behaviors (RB) and Self-Injurious Behaviors (SIB) in Cornelia de Lange Syndrome: A Randomized Double-Blind Placebo-Controlled Pilot Study
Brief Title: Use of N-Acetylcysteine in the Treatment of Repetitive and Self-Injurious Behaviors in Cornelia de Lange Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Cornelia de Lange Syndrome Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00153778
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cornelia de Lange Syndrome
Keywords: Repetitive behaviors; Self-injurious behavior; N-acetylcysteine; Genetic disorder; Children; Psychiatric disease
MeSH Terms: conditions — De Lange Syndrome; Self-Injurious Behavior; Genetic Diseases, Inborn; Mental Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: NAC 1800mg then Placebo (Experimental): NAC 1800 milligrams (mg), oral solution, every 8 hours for 8 weeks, followed by a 2-week wash-out period, followed by NAC Placebo-matching solution, orally every 8 hours, for 8 weeks. Dosage will be titrated weekly starting at 600 mg daily and then increased by 600 mg every week to a target dose of 1800 mg per day.
  Interventions: Drug: N-acetyl cysteine; Other: Placebo
- Group B: Placebo then NAC 1800mg (Experimental): NAC Placebo-matching solution, orally every 8 hours, for 8 weeks, followed by a 2-week wash-out period, followed by NAC 1800 milligrams (mg), oral solution, every 8 hours for 8 weeks. Dosage will be titrated weekly starting at 600 mg daily and then increased by 600 mg every week to a target dose of 1800 mg per day.
  Interventions: Drug: N-acetyl cysteine; Other: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — Oral solution for N-acetyl cysteine is prepared in syringes and provided to the participants along with instructions on how to administer them.
  Other Names: Acetylcysteine; National Drug Code (NDC): 63323-690
Other: Placebo — NAC Placebo-matching solution is prepared in syringes and provided to the participants along with instructions on how to administer them.

SUMMARY:
This research project is a randomized cross-over pilot trial which aims to test the efficacy of N-acetylcysteine (NAC) for the treatment of Repetitive Behaviors (RB) and self-injurious behavior (SIB) in patients with Cornelia de Lange Syndrome (CdLs).

NAC is a known anti-oxidative stress and neuroprotective agent, which has been shown to decrease the occurrence of SIB such as skin picking. NAC has also shown partial response in trials for compulsive behaviors in Obsessive Compulsive Disorder (OCD) and related disorders in autism.

Cornelia de Lange syndrome (CdLS) is a genetic disorder with autistic features, including RBs and SIB. In this randomized clinical trial, participants with CdLS will be blindly assigned one of two possible treatment arms: 1) placebo (8 weeks) and NAC (8 weeks); or 2) NAC (8 weeks) and placebo (8 weeks), with an intermediate 2-week washout period.

DETAILED DESCRIPTION:
Cornelia de Lange syndrome (CdLS) is a genetic condition caused by mutations in cohesin-related genes, mostly notably NIPBL. The CdLS phenotype includes physical features such as typical facies, limb abnormalities, short stature, and hirsutism as well developmental and behavioral manifestations such as intellectual disability, communication deficits, autistic traits and repetitive/self-injurious behaviors (RBs/SIB).

Behavioral challenges such as RBs/SIB pose a significant obstacle to quality of life to individuals with CdLS and families. In CdLS, disruption of developmental systems can impact neuronal and brain development, and impact GABAergic inhibitory interneuron formation, leading to RBs/SIB. Given the potential for dysregulated excitatory glutamatergic output in CdLS, neuronal oxidative stress may play a role in these maladaptive behaviors. NAC replenishes Central Nervous System (CNS) glutathione, a potent antioxidant and may ameliorate RBs/SIB. NAC has been shown to decrease maladaptive behaviors in autism and grooming disorders such as excoriation disorder (skin picking).

An 18-week cross-over trial is proposed to decrease RBs/SIB comprising two 8-week double-blinded active or placebo treatment with a 2-week wash out period in between. A cross-over design will afford for higher efficiency in sample size for similar power. Dosage will be titrated weekly starting at 600 mg daily and then increased by 600 mg every week to a target dose of 1800 mg per day. Participants will be recruited through CdLS Foundation.

Based on a mechanism for regulation glutamate transmission homeostasis in the central nervous system, the use of NAC may be particularly pertinent to individuals with CdLS. It is known that in CdLS genetic networks that impact on limb formation overlap significantly with developmental systems that impact neuronal and brain development, in particular GABAergic inhibitory interneuron formation. Given a dysregulated excitatory glutamatergic mechanism due to interneuron deficits, which can then lead to neuronal oxidative stress and programmed cell death, NAC may act as a key homeostatic regulator to prevent glutamate overactivity and neuronal damage in CdLS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13 to 35 years
* A diagnosis of CdLS as determined by a physician during routine care meeting the major and minor criteria from CdLS guidelines
* Threshold criteria for the presence of RB/SIB as reported on initial screening Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders (CYBOCS-PDD) > 6 OR Aberrant Behavior Checklist (ABC) stereotypy subscale > 7)
* Being able to attend 4 visits over the course of 18 weeks at the Johns Hopkins Hospital
* No acute safety concerns or need for hospitalization due to psychotic, manic or depressive episode
* Not currently pregnant or lactating/breastfeeding. Whether a participant is pregnant or not will be determined by the participant/caregiver report based on date last menses. If there is any suspicion of pregnancy, the PI will confer with the family to obtain testing through the primary care provider.

Exclusion Criteria:

* Allergy to NAC
* Allergy to Quinine
* Contraindication to NAC (organ transplant; untreated or symptomatic gastric condition)
* Need for another medication with which NAC is contraindicated (antibiotics)

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Yale-Brown Obsessive Compulsive Scale Modified for Pervasive Developmental Disorders (CYBOCS-PDD) repetitive behaviors measure score | Baseline, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  CYBOCS-PDD scores range from a minimum of 0 to a maximum of 20, higher scores indicate greater symptom severity. Efficacy of the intervention would be assessed by ≥35% reduction in CYBOCS-PDD repetitive behaviors measure score.
Change in Aberrant Behavior Checklist (ABC) irritability self-injurious behaviors items score | Baseline, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  The ABC irritability sub-scale consists of 15 items of which 3 focus on Self-injurious Behaviors (SIB). Each item takes scores ranging from a minimum of 0 to a maximum of 3. The overall score for the SIB items would range from 0 to 9 with higher scores indicating greater symptom severity. Efficacy of the intervention in reducing self-injurious behaviors would be assessed by a ≥35% reduction in ABC irritability SIB items sub-scale score.

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) irritability non-injurious behaviors items score | Baseline, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  The ABC irritability sub-scale consists of 15 items of which 12 focus on depressed mood and irritable behaviors (non-injurious behaviors). Each item takes a score ranging from a minimum of 0 to a maximum of 3. The overall score for the non-injurious behavior items would range from 0 to 36 with higher scores indicating greater symptom severity. Efficacy of the intervention in reducing depressed mood and irritability would be assessed by a ≥35% score reduction in ABC irritability non-injurious behavior items of sub-scale.
Change in total score of Parenting Stress Index/Short Form (PSI/SF) | Baseline, week 8, week 10, week 18
  The PSI-SF is a 36-item questionnaire designed to measure stress in the parent-child system and identify those families most in need of follow-up services. The PSI-SF consists of three sub-scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Each sub-scale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree). Sub-scale scores therefore range from 12 to 60, whereas the total score ranges from 36 to 180. High scores on the PSI-SF total score indicate greater levels of stress.
Change in Burden Scale for Family Caregivers score | Baseline, week 8, week 10, week 18
  Burden Scale for Family Caregivers, for assessing subjective burden in informal caregivers. It consists of 10 items, each ranging from 0 to 3, with total score ranging from 0 to 30. High scores indicate greater levels of burden in caregiver.
Change in Sensory Profile score | Baseline, week 8, week 10, week 18
  Sensory profile measure identifies sub-types of individuals based on sensory processing patterns and categorize it as one of the following five profiles: 1- Balanced; 2- Interested; 3- Intense; 4- Mellow until ... ; and 5- Vigilant.
Change in Childhood Autism Rating Scale (CARS2) score | Baseline, week 8, week 10, week 18
  The Childhood Autism Rating Scale-Second Edition (CARS2) is a 15-item rating scale used to identify children with autism and distinguishing them from those with developmental disabilities. The 15 items can take 4 scores where 1 stands for normal for child's age, 2 for mildly abnormal, 3 for moderately abnormal and 4 for severely abnormal. Scores range form 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism.
Change in Vineland adaptive Behavior Scale (VABS) score | Baseline, week 8, week 10, week 18
  VABS is a parent interview that provides standard scores (100±15 adjusted for age and gender) for communication, socialization, and daily living.
Change in Clinical Global Impression - Severity of Illness (CGI-S) score | Baseline, week 8, week 10, week 18
  CGI-S asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. Clearly, symptoms and behavior can fluctuate over a week; the score should reflect the average severity level across the seven days.
Change in Side Effects Survey | Baseline, week 2, week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  A previously used side effect tracker is implemented for measuring patient/caregiver-reported side effects of medication. It consists of 14 side effects of interest which each may take scores ranging from 1 defined as "Not reported" through 5 defined as "Disabling".

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Grados, M.D., M.P.H., Principal Investigator — Department of Psychiatry & Behavioral Sciences, Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106